CLINICAL TRIAL: NCT06606457
Title: Pilot of PACE CF, a 3-session Mind-body Pain Management Program for Adults With CF
Brief Title: PACE CF, a 3-session Mind-body Pain Management Program for Adults With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Deborah Friedman, Clinical Psychologist; Assistant Professor of Psychology (Psychiatry), Harvard Medical School; Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024P001312
Record Dates: First submitted 2024-09-10; First posted 2024-09-23 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis (CF); Pain Management
MeSH Terms: conditions — Cystic Fibrosis; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PACE CF Intervention (Experimental): Participants will complete an baseline series of questionnaires, and then meet with the psychologist on their cystic fibrosis care team for 3 weekly meetings to complete the PACE CF program and learn mind-body strategies for pain management. Following completion of the program, they will complete a second assessment that includes another set of questionnaires and a brief qualitative interview to provide feedback about the program.
  Interventions: Behavioral: Pain Acknowledgment Coping and Empowerment in CF (PACE CF)

INTERVENTIONS:
Behavioral: Pain Acknowledgment Coping and Empowerment in CF (PACE CF) — The Pain Acknowledgment Coping and Empowerment in CF (PACE CF) program is a newly developed 3-session mind-body pain management intervention for adults with cystic fibrosis (CF), developed with CF community input. The sessions are delivered by the the CF care team psychologist. Each session will teach mind-body strategies to increase comfort and reduce the impact of pain on the participant's life. These strategies include understanding pain in CF from a mind-body perspective, learning relaxation and mindfulness-based skills, identifying and practicing individualized cognitive and behavioral strategies that improve comfort and well-being, and discussing communication skills that empower people living with CF and pain. Participants will receive a workbook that will provide related education and resources and reinforce skill practice.

SUMMARY:
Many people living with cystic fibrosis (CF) experience pain. However, pain is sometimes unrecognized and under-managed in people with CF. Both medication and non-medication interventions can be used to treat pain and ideally, there is a multicomponent management approach.

The goal of this study is to pilot a new 3-session non-medication mind-body pain management intervention specifically designed for adults with cystic fibrosis (CF). The intervention is titled Pain Acknowledgement Coping and Empowerment in CF (PACE CF).

PACE CF will be administered by a member of the CF care team via telehealth visits to participants at home or during a hospitalization.

The aim of the study is to evaluate the feasibility and patient acceptability of the intervention as well as preliminary evidence of the impact of the intervention on pain and its interference in daily life.

The study will also examine outcomes such as perceived coping, quality of life, symptoms of depression or anxiety, and use of prescribed pain medication, in an exploratory manner.

DETAILED DESCRIPTION:
This study is a multi-center collaboration of a psychological approach to pain treatment in CF. This is the first study to elicit input from the CF community and CF care team members to develop a brief, focused psychological treatment for pain in adults with CF (MGB IRB exempt protocol# 2022P003370). Utilizing the development phase of the grant (protocol# 2022P003370), the investigators developed a brief (3-session) structured intervention manual and patient workbook based on CF community feedback (PACE CF). The intervention will be highly accessible, delivered by a member of the CF care team via telehealth in both inpatient and outpatient settings. The workbook will provide education and resources for patients and reinforce skill practice. Resources will facilitate future training and dissemination, standardization, and evaluation of feasibility, acceptability, and efficacy of the intervention in a larger trial.

The PACE CF intervention integrates the well-established science of behavioral pain management with CF-specific content drawn from feedback from community stakeholders to develop an intervention specific to pain in CF. The investigators anticipate that integration of this intervention into the existing CF model of care will positively impact people with CF by increasing access to best practices in pain treatment, while minimizing additional cost and burden of care.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of CF;
2. age > 18 years;
3. report of pain affecting them at least moderately (score ≥ 2) on the IPOS item;
4. pain lasting at least one month;
5. English-speaking;
6. participant willing and able to give informed consent.

Exclusion Criteria:

Presenting an acute safety risk to self or others at baseline. Participants will not be excluded for the following reasons:

1. CF severity or lung/liver transplant status, if they are otherwise able to participate in CBT;
2. Participation in concomitant pain treatments (e.g., pain medications), as ideally, patients will engage in multi-component pain interventions;
3. psychosocial treatments (with the exception of another formal CBT for pain) or psychopharmacologic treatments at baseline. All concomitant psychosocial and pain-directed treatments will be tracked and considered in analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Acceptability - measured by treatment acceptability interview | End of intervention, up to 2 months
  During visit 5, post-intervention, participants will be asked to complete a brief qualitative interview conducted by a research coordinator regarding treatment acceptability that will be recorded. Interviews will be qualitatively coded utilizing content analysis to summarize feedback regarding intervention acceptability.
Acceptability -Client Satisfaction Questionnaire-8 (CSQ-8) | End of intervention, up to 2 months
  Feedback on the intervention will be obtained from pilot subjects at both sites to assess acceptability of the pain management program.
  At the end of visit 4, after the participant has completed the PACE CF program, participants will complete the Client Satisfaction Questionnaire (CSQ), an 8-item empirically-derived, validated, self-report measure assessing patient satisfaction with health services, rated on a 4-point scale from 1= lowest to 4 = highest satisfaction. The scale has a minimum score of 0, maximum score of 32, with higher scores indicating greater satisfaction.
Feasibility - participant attrition during the intervention period. | From date of baseline assessment to completion of intervention, up to 2 months
  Completion rates will be a key indicator of feasibility. Completion rate will be calculated as the percentage of intervention sessions completed out of the total number of possible sessions (the intervention is 3 sessions) among those enrolled.

SECONDARY OUTCOMES:
Change in pain catastrophizing, measured by the Coping Strategies Questionnaire (CSQ-CAT) | From date of baseline assessment to date of post-intervention assessment, up to 2 months
  This construct will be assessed using the 6-item catastrophizing scale from the Coping Strategies Questionnaire (CSQ-CAT). The catastrophizing scale score ranges from 0 to 36 with higher scores indicating greater pain catastrophizing.
Change in depressive symptoms, measured by the Patient Health Questionnaire-9 (PHQ-9) | From date of baseline assessment to date of post-intervention assessment, up to 2 months
  The Patient Health Questionnaire-9 (PHQ-9) consists of nine questions measuring frequency of depressive symptoms, rated on a Likert scale from 0 "not at all" to 3 ";nearly every day"; with total score ranging 0-27. Clinical severity scores have been established with scores of 5, 10, 15, and 20 representing cut-off scores for mild, moderate, moderately severe, and severe depression, respectively. Higher scores indicate greater clinical severity of depressive symptoms.
Change in anxiety symptoms, measured by the Generalized Anxiety Disorder-7 item scale (GAD-7) | From baseline assessment to post-intervention assessment, up to 2 months
  The Generalized Anxiety Disorder scale (GAD-7) is a 7-item measure of symptoms of anxiety, rated on a Likert scale from 0 "not at all" to 3, "nearly every day", with total scores ranging 0-21. Scores of 5, 10, and 15 correspond to severity ratings of mild, moderate and severe anxiety. Higher scores indicate greater clinical severity of anxiety symptoms.
Change in Health-Related Quality of Life, measured by the Cystic Fibrosis Questionnaire-Revised (CFQ-R) | From baseline assessment to post-intervention assessment, up to 2 months
  The Cystic Fibrosis Questionnaire-Revised (CFQ-R) is a well-established measure of health-related quality of life for people with CF that has been validated in a national, multicenter longitudinal study, demonstrating consistent associations with health outcomes in CF. It consists of 12 scales measuring physical HrQoL (e.g., physical functioning, eating disturbances) or psychosocial HrQoL (e.g., treatment burden, emotional functioning). Each of the 12 scales yield standardized scores ranging from 0 to 100 with higher scores indicating greater health-related quality of life.
Change in sleep quality, measured by the PROMIS Sleep Disturbance Scale short form | From baseline assessment to post-intervention assessment, up to 2 months
  The PROMIS Sleep Disturbance Scale short form (PROMIS SF v1.0 - Sleep Disturbance 6a) is a 6-item validated scale of self-reported perception of sleep quality and disturbance over 7 days. Each item has a 5-point response option. Raw scores range from 6 to 30 and are converted to T-scores, with higher scores indicating greater sleep disturbance.
Change in pain intensity, measured by the PROMIS(r) Pain Intensity Instrument | From date of baseline assessment to date of post-intervention, up to 2 months
  The PROMIS(r) Pain Intensity Instrument (PROMIS Scale v2.0 - Pain Intensity 3a) is a 3- question self-report assessment of pain intensity on a scale from 1 "had no pain" to 5 "very severe." The first 2 questions utilize a 7-day recall and the last question rates pain "right now". Raw summary scores range from 3 to 15, and convert to T-scores, with higher scores indicating greater pain intensity.
Change in pain interference, measured by the PROMIS(r) Pain Interference Scale adult short form | From date of baseline assessment to date of post-intervention assessment, up to 2 months
  The PROMIS(r) Pain Interference Adult Short Form (6 items on a 5-point Likert Scale) measures self-reported consequences of pain on aspects of a person's life. Raw summary scores range from 4 to 20 and convert to T-scores, with higher scores indicating greater pain interference.
Coping Self-Efficacy as measured by the Cystic Fibrosis Coping Self-Efficacy Scale (CF-CSE) | From baseline assessment to post-intervention assessment, up to 2 months
  The Cystic Fibrosis Coping Self-Efficacy Scale was developed by investigators with CF community input. It is a 21-item measure with items rated on a 10-pt scale from "very uncertain" to "very certain," which asks participants to rate their certainty with being able to use a variety of skills and strategies to cope with stress. Some of these strategies reflect core components of CBT; some are specific to coping with CF; many will be targeted in the proposed pain management intervention. The CF Coping Self Efficacy measure contains four subscales: Acceptance/Self-Compassion (4 items), Cognitive Coping/Self-Awareness (8 items), Active Stress Management (4 items) , and Coping with Daily Self-Care Demands (5 items). Higher scores indicated greater coping self-efficacy in each domain of coping skills.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Bruce, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
The study utilizes a small sample and collects mixed method data which may make it difficult to protect the privacy of the participants.